CLINICAL TRIAL: NCT01049789
Title: Treatment for Depression Among HIV-Infected Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATN 080
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-03

CONDITIONS: HIV; Depression; HIV Infections
Keywords: youth; HIV; Depression; Cognitive Behavioral Therapy; Medication management
MeSH Terms: conditions — Depression; HIV Infections | interventions — Cognitive Behavioral Therapy; Medication Therapy Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAU (Active Comparator): Sites participating in Phase I and Phase II will be randomized to implement this treatment method or the other treatment method. All ATN 080 participants at a site randomized to implement TAU will receive that treatment method.
  Interventions: Behavioral: TAU - Treatment as Usual
- COMB (Experimental): Sites participating in Phase I and Phase II will be randomized to implement this treatment method or the other treatment method. All ATN 080 participants at a site randomized to implement COMB will receive that treatment method.
  Interventions: Behavioral: COMB - Combination Cognitive Behavioral Therapy and Medication Management

INTERVENTIONS:
Behavioral: COMB - Combination Cognitive Behavioral Therapy and Medication Management — Phase I: 24-week intervention consisting of Cognitive Behavioral Therapy (CBT) and Medication Management (MM) manuals. Study coordinators and site clinicians will document depression symptoms and treatment regimens for all participants for 24 weeks. Site staff and participants at COMB sites will participate in an exit interview and findings will be used to revise CBT and MM intervention manuals at the end of Phase I.
  Phase II: similar procedures as Phase I; COMB sites will implement the revised CBT and MM manuals. Depression symptoms and treatment regimens for all participants will be documented for 24 weeks. All Phase II participants will have 2 follow-up visits at weeks 36 and 48.
  Other Names: Cognitive Behavioral Therapy (CBT); Medication Management (MM)
  Arms: COMB
Behavioral: TAU - Treatment as Usual — Phase I: Participants enrolled at TAU sites will receive treatment for depression that is typical at that site, which may include medication management, psychosocial therapy, or a combination of the two.
  Phase II: Participants at TAU sites will receive treatment for depression that is typical at that site. As in Phase I, psychopharmacological and psychosocial interventions will not be standardized and participants may receive any depression treatment recommended by the site clinicians while on study. Depression symptoms and treatment regimens for all participants will be documented for 24 weeks. Additionally, all Phase II participants will have 2 follow-up visits at weeks 36 and 48.
  Arms: TAU

SUMMARY:
This is a two-phase study that is designed to test a novel behavioral intervention to treat depression in Human Immunodeficiency Virus (HIV) adolescents and young adults. Four Adolescent Trials Network (ATN) sites will be assigned to either the Combination Cognitive Behavioral Therapy and Medication Management (COMB) treatment group or the Treatment as Usual (TAU) group.

Phase I involves pilot testing of a 24-week intervention consisting of Cognitive Behavioral Therapy (CBT) and Medication Management (MM) manuals at sites assigned to the COMB treatment group. Participants enrolled at TAU sites will receive treatment for depression that is typical at that site, which may include medication management, psychosocial therapy, or a combination of the two. Psychopharmacological and psychosocial interventions will not be standardized and participants may receive any depression treatment recommended by the site clinicians while on study. Study coordinators and site clinicians, regardless of group assignment, will document depression symptoms and treatment regimens for all participants for 24 weeks. In addition, site staff and participants at COMB sites will participate in an exit interview. The findings from these interviews will be used to revise both CBT and MM intervention manuals at the end of Phase I.

Phase II is a feasibility study of the revised CBT and MM manuals. Phase II involves similar procedures as Phase I; sites assigned to COMB will implement the revised CBT and MM manuals. Participants at TAU sites will receive treatment for depression that is typical at that site. As in Phase I, psychopharmacological and psychosocial interventions will not be standardized and participants may receive any depression treatment recommended by the site clinicians while on study. Depression symptoms and treatment regimens for all participants will be documented for 24 weeks. Additionally, all Phase II participants will have 2 follow-up visits at weeks 36 and 48. Again, site staff and participants at COMB sites will participate in an exit interview. The findings from these interviews will be used to revise both CBT and MM manuals at the end of Phase II.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults ages 16 years and 0 days to 24 years and 364 days at time of enrollment;
* Engaged in care at the participating AMTU;
* Documented HIV infection by medical record review or verbal verification from referring professional and aware of their HIV status;
* Primary diagnosis of non-psychotic depression, either MDD, Depression NOS, or Dysthymia, as defined by DSM-IV criteria and as documented prior to study screening by treating licensed mental health clinician;
* Current depressive symptoms warranting intervention as determined by treating licensed mental health clinician with a score of ≥ 7 on the QIDS-C; NOTE: Youth already receiving treatment for depression with QIDS-C scores ≥ 7 are eligible but those with scores < 7, indicating who minimal ongoing depressive symptoms, are not eligible.
* Ability to understand written and spoken English; and
* Ability and willingness to provide informed consent or assent.

Exclusion Criteria:

* Known or self-reported by participant to have a history of any psychotic disorder (including depression with psychotic features) and/or bipolar I or II disorder;
* Alcohol or substance dependence based on DSM-IV criteria within the past six months as determined by treating licensed mental health clinician. Any cases that are uncertain require Protocol Team approval;
* Pregnant or breast-feeding females;
* Known or self-reported by participant (or parent if available) to have a first degree relative(s) with Bipolar I Disorder;
* Depression and/or suicidal ideation requiring more intensive treatment than the study provides or at immediate risk of being a danger to themselves or others as determined by treating licensed mental health clinician;
* Cognitive limitations, emotional instability or medical illness as determined by treating licensed mental health clinician and/or study coordinator; and
* For Phase II only, previous participation in Phase I.
* For participants at COMB sites only, ongoing CBT for treatment of depressive symptoms at time of study enrollment (e.g., teaching cognitive restructuring using role-play, identification of cognitive distortions, automatic thoughts, dysfunctional attitudes); and NOTE: Youth who received CBT in the past may be considered for enrollment. Any cases that are uncertain require Protocol Team approval.
* For participants at COMB sites only, continuing antidepressant management by a site clinician who is not trained in COMB.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2010-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Ph. I: To pilot manuals for CBT and MM for treatment of depression in people ages 16-24 infected with HIV that target symptoms of depression, and motivation for medical and depression treatment, adherence to medical care and wellness behaviors. | 1 year
Ph I and II: To examine acceptability of study participation, feasibility of participation in such a study and participant satisfaction with the intervention | 3 years
Ph I: To examine the feasibility of collecting depression treatment data as well as data from other desired outcome measures at COMB and TAU sites. | 1 year
Ph I and II: To revise the manuals based on feedback received in the Phase I from participants, providers and the examination of analyses of adherence and depressive symptom outcomes. | 3 years
Ph II: To examine whether participants receiving COMB have improved depression and medical treatment adherence (e.g., more kept medical and mental health visits, fewer treatment dropouts) compared to participants receiving TAU. | 2 years
Ph II: To examine whether participants receiving COMB demonstrate improved depression outcomes (e.g., decreased depressive symptoms, greater remission rates, and decreased relapse rates) compared to the TAU condition. | 2 years

SECONDARY OUTCOMES:
Ph I: To examine whether participants receiving COMB) have improved depression and medical treatment adherence (e.g., more kept medical and mental health visits, fewer treatment dropouts) compared to participants receiving TAU. | 1 year
Ph I: To examine whether participants receiving COMB demonstrate improved depression outcomes (e.g., decreased depressive symptoms, greater remission rates, and decreased relapse rates) compared to participants receiving TAU. | 1 year
Ph II: Examine whether participants receiving COMB demonstrate improved medical outcomes (e.g., increased CD4 T-cell count, decreased HIV Ribonucleic Acid (RNA) level). | 2 years
Ph II: Obtain preliminary descriptive data on what TAU consists of for participants with HIV and depression in this age group. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Larry Brown, MD, Study Chair — Adolescent Trials Network
Locations (4):
- United States (4):
  - USF College of Medicine, Tampa, Florida
  - Montefiore Medical Center, The Bronx, New York
  - The Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Center, Memphis, Tennessee

REFERENCES:
- See also: ATN Website — http://www.atnonline.org